CLINICAL TRIAL: NCT06904976
Title: Nature-Focused Mindfulness and Spiritual Well-being Among Adults with Moderate Prolonged Grief Symptoms: a Randomized Controlled Trial
Brief Title: Nature-Focused Mindfulness and Spiritual Well-being Among Adults with Moderate Prolonged Grief Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Twente (Other)
Responsible Party: Principal Investigator, Jannis Kraiss, Principal Investigator, University of Twente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 250441
Record Dates: First submitted 2025-03-12; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Grief; Spiritual Wellbeing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nature-focused mindfulness (Experimental): 10 minutes walking to a chosen natural location, 10 minutes guided mindfulness practice, 10 minutes walking back.
  Interventions: Behavioral: Nature-focused mindfulness
- Noticing-nature (Active Comparator): walk in nature for 30 minutes per day and pay attention to how the natural objects/scenes they encounter in their daily surroundings make them feel over the 14-day period.
  Interventions: Behavioral: Noticing-nature
- Waitlist (No Intervention)

INTERVENTIONS:
Behavioral: Nature-focused mindfulness — The intervention consisted of a daily 30-minute self-guided practice structured in three parts: (1) participants first walked mindfully for 10 minutes in a natural environment of their choosing (e.g., local park, forest, garden), (2) upon reaching a suitable location, they engaged in a 10-minute guided mindfulness practice, and (3) concluded with a 10-minute mindful walk back.
  Arms: Nature-focused mindfulness
Behavioral: Noticing-nature — Participants allocated to the noticing-nature active control group will be instructed to walk in nature for 30 minutes per day and pay attention to how the natural objects/scenes they encounter in their daily surroundings make them feel over the 14-day period.
  Arms: Noticing-nature

SUMMARY:
The goal of this randomized controlled trial is to evaluate whether a nature-focused mindfulness intervention can enhance spiritual well-being and reduce grief symptoms among adults with moderate prolonged grief symptoms. The main questions it aims to answer are:

Does a nature-focused mindfulness intervention improve spiritual well-being compared to an active control condition (noticing nature) and a waitlist control condition?

Does a nature-focused mindfulness intervention reduce grief severity and improve mental well-being, nature connectedness, selflessness, ability to adapt, personal recovery, and elevation compared to control conditions?

How do spiritual well-being, ability to adapt, nature connectedness, selflessness, grief reactions, and positive/negative affect change during the intervention period?

Researchers will compare a nature-focused mindfulness intervention to both a noticing-nature active control group and a waitlist control group to isolate mindfulness-specific effects from possible general nature exposure benefits.

Participants will:

Complete baseline, post-intervention, and follow-up assessments (at one and three months) Engage in either 10 sessions of nature-focused mindfulness practice or noticing nature activities over a two-week period (intervention and active control groups) Provide daily diary responses about their experiences throughout the 14-day intervention period

ELIGIBILITY:
Inclusion Criteria:

* Be a family member, spouse, or friend of a person who died at least 6 months prior to study enrollment;
* Be ≥18 years of age;
* Report moderate subclinical grief (score range from 47-70) based on the Traumatic Grief Inventory-Self Report Plus (TGI-SR+, Lenferink, Eisma, et al., 2022);
* Have access to a natural environment suitable for the intervention;
* Be willing and able to move in nature daily (with or without mobility assistance devices) and engage in brief mindfulness practices;
* Have sufficient Dutch language proficiency;
* Have access to Internet and mobile applications.

Exclusion Criteria:

* Acute suicide risk assessed in the screening step;
* A score lower than 47 or higher than 70 on TGI-SR+;
* Physical limitations that prevent moving outdoors for 30 minutes daily, even with mobility assistance devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-03-24 (Estimated); Primary Completion 2025-09-09 (Estimated); Study Completion 2025-09-09 (Estimated)

PRIMARY OUTCOMES:
Spiritual well-being measured by Spiritual Attitude and Involvement List-Short Form | Baseline
  Measured using the Spiritual Attitude and Involvement List-Short Form (SAIL-SF; Bohlmeijer et al., 2023). The SAIL-SF measures seven dimensions of spiritual well-being: meaningfulness, trust, acceptance, caring for others, connectedness with nature, transcendent experiences, and spiritual activities. Each dimension is assessed by one item (e.g., "I experience the things I do as meaningful", "I try to take life as it comes"). Items are rated on a 6-point Likert scale ranging from 1 (not at all) to 6 (to a very high degree), with higher scores indicating greater spiritual well-being. The total score is calculated as the mean of all items.
Spiritual well-being measured by Spiritual Attitude and Involvement List-Short Form | 1 month after baseline
  Measured using the Spiritual Attitude and Involvement List-Short Form (SAIL-SF; Bohlmeijer et al., 2023). The SAIL-SF measures seven dimensions of spiritual well-being: meaningfulness, trust, acceptance, caring for others, connectedness with nature, transcendent experiences, and spiritual activities. Each dimension is assessed by one item (e.g., "I experience the things I do as meaningful", "I try to take life as it comes"). Items are rated on a 6-point Likert scale ranging from 1 (not at all) to 6 (to a very high degree), with higher scores indicating greater spiritual well-being. The total score is calculated as the mean of all items.
Spiritual well-being measured by Spiritual Attitude and Involvement List-Short Form | 2 months after baseline
  Measured using the Spiritual Attitude and Involvement List-Short Form (SAIL-SF; Bohlmeijer et al., 2023). The SAIL-SF measures seven dimensions of spiritual well-being: meaningfulness, trust, acceptance, caring for others, connectedness with nature, transcendent experiences, and spiritual activities. Each dimension is assessed by one item (e.g., "I experience the things I do as meaningful", "I try to take life as it comes"). Items are rated on a 6-point Likert scale ranging from 1 (not at all) to 6 (to a very high degree), with higher scores indicating greater spiritual well-being. The total score is calculated as the mean of all items.
Spiritual well-being measured by Spiritual Attitude and Involvement List-Short Form | 4 months after baseline
  Measured using the Spiritual Attitude and Involvement List-Short Form (SAIL-SF; Bohlmeijer et al., 2023). The SAIL-SF measures seven dimensions of spiritual well-being: meaningfulness, trust, acceptance, caring for others, connectedness with nature, transcendent experiences, and spiritual activities. Each dimension is assessed by one item (e.g., "I experience the things I do as meaningful", "I try to take life as it comes"). Items are rated on a 6-point Likert scale ranging from 1 (not at all) to 6 (to a very high degree), with higher scores indicating greater spiritual well-being. The total score is calculated as the mean of all items.

SECONDARY OUTCOMES:
Grief intensity measured by Traumatic Grief Inventory-Self Report Plus | Baseline
  Measured using the 22-item Traumatic Grief Inventory-Self Report Plus (TGI-SR+; Lenferink et al., 2022). Participants rated the extent to which they experienced each grief symptom during the past two weeks on 5-point Likert scale (1 = never to 5 = always). Total scores are calculated by summing all items (range: 22-110), with higher scores indicating greater grief intensity. A total score ≥71 indicates probable clinical DSM-5-TR PGD.
Grief intensity measured by Traumatic Grief Inventory-Self Report Plus | 1 month after baseline
  Measured using the 22-item Traumatic Grief Inventory-Self Report Plus (TGI-SR+; Lenferink et al., 2022). Participants rated the extent to which they experienced each grief symptom during the past two weeks on 5-point Likert scale (1 = never to 5 = always). Total scores are calculated by summing all items (range: 22-110), with higher scores indicating greater grief intensity. A total score ≥71 indicates probable clinical DSM-5-TR PGD.
Grief intensity measured by Traumatic Grief Inventory-Self Report Plus | 2 months after baseline
  Measured using the 22-item Traumatic Grief Inventory-Self Report Plus (TGI-SR+; Lenferink et al., 2022). Participants rated the extent to which they experienced each grief symptom during the past two weeks on 5-point Likert scale (1 = never to 5 = always). Total scores are calculated by summing all items (range: 22-110), with higher scores indicating greater grief intensity. A total score ≥71 indicates probable clinical DSM-5-TR PGD.
Grief intensity measured by Traumatic Grief Inventory-Self Report Plus | 4 months after baseline
  Measured using the 22-item Traumatic Grief Inventory-Self Report Plus (TGI-SR+; Lenferink et al., 2022). Participants rated the extent to which they experienced each grief symptom during the past two weeks on 5-point Likert scale (1 = never to 5 = always). Total scores are calculated by summing all items (range: 22-110), with higher scores indicating greater grief intensity. A total score ≥71 indicates probable clinical DSM-5-TR PGD.
Nature connectedness measured by Inclusion of Nature in Self scale | Baseline
  Measured using 1-item Inclusion of Nature in Self scale (INS; Schultz, 2001). The INS is a single-item pictorial measure that assesses the extent to which individuals include nature within their cognitive representation of self. The measure consists of seven pairs of circles labeled "self" and "nature" with varying degrees of overlap, from completely separate (1) to almost completely overlapping (7). Participants select the picture that best describes their relationship with the natural environment.
Nature connectedness measured by Inclusion of Nature in Self scale | 1 month after baseline
  Measured using 1-item Inclusion of Nature in Self scale (INS; Schultz, 2001). The INS is a single-item pictorial measure that assesses the extent to which individuals include nature within their cognitive representation of self. The measure consists of seven pairs of circles labeled "self" and "nature" with varying degrees of overlap, from completely separate (1) to almost completely overlapping (7). Participants select the picture that best describes their relationship with the natural environment.
Nature connectedness measured by Inclusion of Nature in Self scale | 2 months after baseline
  Measured using 1-item Inclusion of Nature in Self scale (INS; Schultz, 2001). The INS is a single-item pictorial measure that assesses the extent to which individuals include nature within their cognitive representation of self. The measure consists of seven pairs of circles labeled "self" and "nature" with varying degrees of overlap, from completely separate (1) to almost completely overlapping (7). Participants select the picture that best describes their relationship with the natural environment.
Nature connectedness measured by Inclusion of Nature in Self scale | 4 months after baseline
  Measured using 1-item Inclusion of Nature in Self scale (INS; Schultz, 2001). The INS is a single-item pictorial measure that assesses the extent to which individuals include nature within their cognitive representation of self. The measure consists of seven pairs of circles labeled "self" and "nature" with varying degrees of overlap, from completely separate (1) to almost completely overlapping (7). Participants select the picture that best describes their relationship with the natural environment.
Nature connectedness measured by Connectedness to Nature Scale | Baseline
  Measured using 14-item Connectedness to Nature Scale (CNS; Mayer & Frantz, 2004). The CNS measures individuals' trait levels of feeling emotionally and experientially connected to the natural world. Participants rated items such as "I often feel a sense of oneness with the natural world around me" and "I think of the natural world as a community to which I belong" on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). The total score is calculated as the mean of all items after reverse-scoring items 4, 12, and 14, with higher scores indicating greater connectedness to nature.
Nature connectedness measured by Connectedness to Nature Scale | 1 month after baseline
  Measured using 14-item Connectedness to Nature Scale (CNS; Mayer & Frantz, 2004). The CNS measures individuals' trait levels of feeling emotionally and experientially connected to the natural world. Participants rated items such as "I often feel a sense of oneness with the natural world around me" and "I think of the natural world as a community to which I belong" on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). The total score is calculated as the mean of all items after reverse-scoring items 4, 12, and 14, with higher scores indicating greater connectedness to nature.
Nature connectedness measured by Connectedness to Nature Scale | 2 months after baseline
  Measured using 14-item Connectedness to Nature Scale (CNS; Mayer & Frantz, 2004). The CNS measures individuals' trait levels of feeling emotionally and experientially connected to the natural world. Participants rated items such as "I often feel a sense of oneness with the natural world around me" and "I think of the natural world as a community to which I belong" on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). The total score is calculated as the mean of all items after reverse-scoring items 4, 12, and 14, with higher scores indicating greater connectedness to nature.
Nature connectedness measured by Connectedness to Nature Scale | 4 months after baseline
  Measured using 14-item Connectedness to Nature Scale (CNS; Mayer & Frantz, 2004). The CNS measures individuals' trait levels of feeling emotionally and experientially connected to the natural world. Participants rated items such as "I often feel a sense of oneness with the natural world around me" and "I think of the natural world as a community to which I belong" on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). The total score is calculated as the mean of all items after reverse-scoring items 4, 12, and 14, with higher scores indicating greater connectedness to nature.
Mental well-being measured by Mental Health Continuum-Short Form | Baseline
  Measured using the Mental Health Continuum-Short Form (MHC-SF; Lamers et al., 2011), a 14-item scale measuring three dimensions of well-being: emotional (3 items), psychological (6 items), and social well-being (5 items). Participants rated the frequency of experiencing various feelings of well-being during the past month on a 6-point Likert scale (0 = never to 5 = every day). Scores are calculated as the mean of all items, with higher scores indicating greater well-being.
Mental well-being measured by Mental Health Continuum-Short Form | 1 month after baseline
  Measured using the Mental Health Continuum-Short Form (MHC-SF; Lamers et al., 2011), a 14-item scale measuring three dimensions of well-being: emotional (3 items), psychological (6 items), and social well-being (5 items). Participants rated the frequency of experiencing various feelings of well-being during the past month on a 6-point Likert scale (0 = never to 5 = every day). Scores are calculated as the mean of all items, with higher scores indicating greater well-being.
Mental well-being measured by Mental Health Continuum-Short Form | 2 months after baseline
  Measured using the Mental Health Continuum-Short Form (MHC-SF; Lamers et al., 2011), a 14-item scale measuring three dimensions of well-being: emotional (3 items), psychological (6 items), and social well-being (5 items). Participants rated the frequency of experiencing various feelings of well-being during the past month on a 6-point Likert scale (0 = never to 5 = every day). Scores are calculated as the mean of all items, with higher scores indicating greater well-being.
Mental well-being measured by Mental Health Continuum-Short Form | 4 months after baseline
  Measured using the Mental Health Continuum-Short Form (MHC-SF; Lamers et al., 2011), a 14-item scale measuring three dimensions of well-being: emotional (3 items), psychological (6 items), and social well-being (5 items). Participants rated the frequency of experiencing various feelings of well-being during the past month on a 6-point Likert scale (0 = never to 5 = every day). Scores are calculated as the mean of all items, with higher scores indicating greater well-being.
Selflessness measured by Perceived Body Boundaries Scale | Baseline
  Perceived Body Boundaries Scale (PBBS; Dambrun, 2016). This scale comprises a single item designed to assess the strength of participants' perceived body boundaries.
  A series of images of human forms with increasingly transparent boundaries to indicate gradations of body boundary salience. "Which images best represent your perception of your body's boundaries right now?" Responses range from 1 (no boundary dissolution) to 7 (a lot of boundary dissolution).
Selflessness measured by Perceived Body Boundaries Scale | 1 month after baseline
  Perceived Body Boundaries Scale (PBBS; Dambrun, 2016). This scale comprises a single item designed to assess the strength of participants' perceived body boundaries.
  A series of images of human forms with increasingly transparent boundaries to indicate gradations of body boundary salience. "Which images best represent your perception of your body's boundaries right now?" Responses range from 1 (no boundary dissolution) to 7 (a lot of boundary dissolution).
Selflessness measured by Perceived Body Boundaries Scale | 2 months after baseline
  Perceived Body Boundaries Scale (PBBS; Dambrun, 2016). This scale comprises a single item designed to assess the strength of participants' perceived body boundaries.
  A series of images of human forms with increasingly transparent boundaries to indicate gradations of body boundary salience. "Which images best represent your perception of your body's boundaries right now?" Responses range from 1 (no boundary dissolution) to 7 (a lot of boundary dissolution).
Selflessness measured by Perceived Body Boundaries Scale | 4 months after baseline
  Perceived Body Boundaries Scale (PBBS; Dambrun, 2016). This scale comprises a single item designed to assess the strength of participants' perceived body boundaries.
  A series of images of human forms with increasingly transparent boundaries to indicate gradations of body boundary salience. "Which images best represent your perception of your body's boundaries right now?" Responses range from 1 (no boundary dissolution) to 7 (a lot of boundary dissolution).
Selflessness measured by Spatial Frame of Reference Continuum | Baseline
  Spatial Frame of Reference Continuum (SFoRC; Hanley & Garland, 2019). This scale comprises a single item used to assess the extent to which the field of awareness is perceived to extend beyond the physical body.
  How far does your self extend into the world? Using the letters and image below, please indicate how far you feel that your self extends beyond your physical body. "A" represents your self stopping at your physical body. "F" represents your self extending into everything (e.g., the entire Universe). The letters inbetween "A" and "F" represent different levels of self-extension. The rings are symbolic, and do not represent actual distances.
Selflessness (Spatial Frame of Reference Continuum) | 1 month after baseline
  Spatial Frame of Reference Continuum (SFoRC; Hanley & Garland, 2019). This scale comprises a single item used to assess the extent to which the field of awareness is perceived to extend beyond the physical body.
  How far does your self extend into the world? Using the letters and image below, please indicate how far you feel that your self extends beyond your physical body. "A" represents your self stopping at your physical body. "F" represents your self extending into everything (e.g., the entire Universe). The letters inbetween "A" and "F" represent different levels of self-extension. The rings are symbolic, and do not represent actual distances.
Selflessness measured by Spatial Frame of Reference Continuum | 2 months after baseline
  Spatial Frame of Reference Continuum (SFoRC; Hanley & Garland, 2019). This scale comprises a single item used to assess the extent to which the field of awareness is perceived to extend beyond the physical body.
  How far does your self extend into the world? Using the letters and image below, please indicate how far you feel that your self extends beyond your physical body. "A" represents your self stopping at your physical body. "F" represents your self extending into everything (e.g., the entire Universe). The letters inbetween "A" and "F" represent different levels of self-extension. The rings are symbolic, and do not represent actual distances.
Selflessness measured by Spatial Frame of Reference Continuum | 4 months after baseline
  Spatial Frame of Reference Continuum (SFoRC; Hanley & Garland, 2019). This scale comprises a single item used to assess the extent to which the field of awareness is perceived to extend beyond the physical body.
  How far does your self extend into the world? Using the letters and image below, please indicate how far you feel that your self extends beyond your physical body. "A" represents your self stopping at your physical body. "F" represents your self extending into everything (e.g., the entire Universe). The letters inbetween "A" and "F" represent different levels of self-extension. The rings are symbolic, and do not represent actual distances.
Elevation measured by Elevating Experiences Scale | Baseline
  Measured using the Elevating Experiences Scale (EES; Huta & Ryan, 2010), a 13-item measure that captures feelings of transcendence, moral inspiration, and connection to something greater than oneself. Participants rated their experiences over the past two weeks using a 7-point Likert-type scale ranging from 1 (not at all) to 7 (extremely). Scores are calculated as the mean of all items, with higher scores indicating greater elevation.
Elevation measured by Elevating Experiences Scale | 1 month after baseline
  Measured using the Elevating Experiences Scale (EES; Huta & Ryan, 2010), a 13-item measure that captures feelings of transcendence, moral inspiration, and connection to something greater than oneself. Participants rated their experiences over the past two weeks using a 7-point Likert-type scale ranging from 1 (not at all) to 7 (extremely). Scores are calculated as the mean of all items, with higher scores indicating greater elevation.
Elevation measured by Elevating Experiences Scale | 2 months after baseline
  Measured using the Elevating Experiences Scale (EES; Huta & Ryan, 2010), a 13-item measure that captures feelings of transcendence, moral inspiration, and connection to something greater than oneself. Participants rated their experiences over the past two weeks using a 7-point Likert-type scale ranging from 1 (not at all) to 7 (extremely). Scores are calculated as the mean of all items, with higher scores indicating greater elevation.
Elevation measured by Elevating Experiences Scale | 4 months after baseline
  Measured using the Elevating Experiences Scale (EES; Huta & Ryan, 2010), a 13-item measure that captures feelings of transcendence, moral inspiration, and connection to something greater than oneself. Participants rated their experiences over the past two weeks using a 7-point Likert-type scale ranging from 1 (not at all) to 7 (extremely). Scores are calculated as the mean of all items, with higher scores indicating greater elevation.
Ability to adapt measured by Generic Sense of Ability to Adapt Scale | Baseline
  Measured using the Generic Sense of Ability to Adapt Scale (GSAAS; Franken et al., 2023). The GSAAS is a 10-item scale measuring perceived ability to readjust and actively deal with the psychosocial consequences of challenging events. Items (e.g., "If something unexpected happens, I can easily adapt") are rated on a 5-point Likert scale from "not at all" (0) to "always" (4). The total score is calculated as the mean of all items, with higher scores indicating greater ability to adapt.
Ability to adapt measured by Generic Sense of Ability to Adapt Scale | 1 month after baseline
  Measured using the Generic Sense of Ability to Adapt Scale (GSAAS; Franken et al., 2023). The GSAAS is a 10-item scale measuring perceived ability to readjust and actively deal with the psychosocial consequences of challenging events. Items (e.g., "If something unexpected happens, I can easily adapt") are rated on a 5-point Likert scale from "not at all" (0) to "always" (4). The total score is calculated as the mean of all items, with higher scores indicating greater ability to adapt.
Ability to adapt measured by Generic Sense of Ability to Adapt Scale | 2 months after baseline
  Measured using the Generic Sense of Ability to Adapt Scale (GSAAS; Franken et al., 2023). The GSAAS is a 10-item scale measuring perceived ability to readjust and actively deal with the psychosocial consequences of challenging events. Items (e.g., "If something unexpected happens, I can easily adapt") are rated on a 5-point Likert scale from "not at all" (0) to "always" (4). The total score is calculated as the mean of all items, with higher scores indicating greater ability to adapt.
Ability to adapt measured by Generic Sense of Ability to Adapt Scale | 4 months after baseline
  Measured using the Generic Sense of Ability to Adapt Scale (GSAAS; Franken et al., 2023). The GSAAS is a 10-item scale measuring perceived ability to readjust and actively deal with the psychosocial consequences of challenging events. Items (e.g., "If something unexpected happens, I can easily adapt") are rated on a 5-point Likert scale from "not at all" (0) to "always" (4). The total score is calculated as the mean of all items, with higher scores indicating greater ability to adapt.
Personal recovery measured by Brief INSPIRE-O | Baseline
  Measured using the 5-item Brief INSPIRE-O, modified from the Brief INSPIRE support measure (Williams et al., 2015). Items are rated on a 5-point Likert scale from 0 (not at all) to 4 (very much). Following scoring guidelines (Moeller et al., 2023), raw scores were summed and multiplied by 5 to give a total score ranging from 0 to 100, with higher scores indicating better personal functioning.
Personal recovery measured by Brief INSPIRE-O | 1 month after baseline
  Measured using the 5-item Brief INSPIRE-O, modified from the Brief INSPIRE support measure (Williams et al., 2015). Items are rated on a 5-point Likert scale from 0 (not at all) to 4 (very much). Following scoring guidelines (Moeller et al., 2023), raw scores were summed and multiplied by 5 to give a total score ranging from 0 to 100, with higher scores indicating better personal functioning.
Personal recovery measured by Brief INSPIRE-O | 2 months after baseline
  Measured using the 5-item Brief INSPIRE-O, modified from the Brief INSPIRE support measure (Williams et al., 2015). Items are rated on a 5-point Likert scale from 0 (not at all) to 4 (very much). Following scoring guidelines (Moeller et al., 2023), raw scores were summed and multiplied by 5 to give a total score ranging from 0 to 100, with higher scores indicating better personal functioning.
Personal recovery measured by Brief INSPIRE-O | 4 months after baseline
  Measured using the 5-item Brief INSPIRE-O, modified from the Brief INSPIRE support measure (Williams et al., 2015). Items are rated on a 5-point Likert scale from 0 (not at all) to 4 (very much). Following scoring guidelines (Moeller et al., 2023), raw scores were summed and multiplied by 5 to give a total score ranging from 0 to 100, with higher scores indicating better personal functioning.
Daily diary (assessed daily during 14-day intervention period) | From baseline to post-intervention (2-weeks)
  "Please respond to the following items based on your experiences and feelings today, reflecting specifically on the past 24 hours." Responses range from 1 (not at all) to 7 (very much).
  1. Grief reactions (2 items)
  2. Positive affect (2 items)
  3. Negative affect (2 items)
  4. Nature connectedness (1 item; Schultz, 2001)
  5. Selflessness (1 item; Dambrun, 2016)
  6. Spiritual well-being (1 item; Underwood, 2011)
  7. Ability to adapt (1 item; Franken et al., 2023)
     * Analysis metric: Daily fluctuations and sudden gains

OTHER OUTCOMES:
Demographic characteristics | Baseline
  Age, gender, education level, employment status
Loss-related characteristics | Baseline
  (1) Relationship to the deceased (categorized as spouse/partner, child, parent, sibling, other family member, or friend); (2) Time since loss (measured in months since death occurred); and (3) Cause of death (categorized as natural anticipated, natural sudden, accident, suicide, homicide, or other/unknown). These variables will be reported using descriptive statistics, with categorical variables presented as frequencies and percentages, and continuous variables (time since loss) presented as means and standard deviations.
Previous mindfulness experience | Baseline
  Using two complementary items. First, participants will respond to the question "Do you have experience with meditation?" with three response options: "Yes, I would call myself an expert and have a lot of experience with meditation," "Yes, I have a little experience with meditation," or "No, I have no experience with meditation (yet)." Second, current practice frequency will be assessed with the question "How many times have you meditated in the past month?" with four response options: "Daily," "Weekly," "Occasionally," or "Never."
Previous Nature experience | Baseline
  Participants will respond to the question "Are you regularly in nature (such as the forest, a park or the beach)?" with five response options: "Yes, every day," "Yes, one or more times a week," "Yes, once a month," "No, rarely," or "No, never."
Intervention adherence | 1 month after baseline
  A post-intervention adherence item measuring self-reported frequency of practice completion and duration of practice sessions. Adherence will be operationalized as the percentage of assigned sessions completed (ranging from 0-100%) and reported as means, standard deviations, and frequency distributions.
Co-intervention use | 1 month after baseline
  Participants will respond to the question: "During the past 2 weeks, did you receive additional psychological professional support from a psychologist, therapist, or psychiatrist for dealing with your emotional problems?" Results will be reported as frequencies and percentages. Co-intervention use will be examined as a potential confounding variable in the analysis to determine whether concurrent psychological support interacts with the intervention effects.
Client satisfaction measured by Client Satisfaction Questionnaire | 1 month after baseline
  Measured using 8-item Client Satisfaction Questionnaire (CSQ-8; Attkisson & Zwick, 1982). Items will be scored on a 4-point scale, and a sum score (8-32) will be calculated with higher scores being indicative of a larger satisfaction with the intervention.

IPD SHARING:
Plan to Share IPD: Undecided